CLINICAL TRIAL: NCT01186783
Title: Reducing Elevated Heart Rate in Patients With Multiple Organ Dysfunction Syndrome (MODS) by the "Funny Channel" Current (If) Inhibitor Ivabradine
Brief Title: Reducing Elevated Heart Rate in Patients With Multiple Organ Dysfunction Syndrome (MODS) by Ivabradine
Acronym: MODIfY
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: Servier (Industry); KKS Netzwerk (Network)
Responsible Party: Karl Werdan, MD, Professor, Medical Faculty of the Martin-Luther-University Halle-Wittenberg, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KKSH-067
Record Dates: First submitted 2010-08-17; First posted 2010-08-23 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Multiple Organ Dysfunction Syndrome
Keywords: heart rate; multiple organ dysfunction syndrome; ivabradine; sepsis; cardiogenic shock
MeSH Terms: conditions — Multiple Organ Failure; Sepsis; Shock, Cardiogenic | interventions — Ivabradine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard treatment (No Intervention): All patients receive established medical therapy according to current guidelines and therapeutic standards.
- ivabradine (add-on) (Active Comparator): Patients in the ivabradine treatment arm receive an additional enteral preparation (orally, via nasogastric tube or percutaneous endoscopic gastrostomy-probe) of ivabradine for 4 days.
  Interventions: Drug: ivabradine

INTERVENTIONS:
Drug: ivabradine — Patients in the ivabradine treatment arm receive an additional enteral preparation (orally, via nasogastric tube or percutaneous endoscopic gastrostomy-probe) of ivabradine for 4 days.
  Day 1 and 2:
  5,0 mg ivabradine b.i.d. if heart rate ≥60bpm (acute renal failure: ≥70bpm)
  Day 3 and 4:
  5,0 mg ivabradine b.i.d. if 60bpm≥heart rate<90bpm (acute renal failure: 70bpm≥heart rate <90bpm
  7,5 mg ivabradine b.i.d. if heart rate ≥90bpm
  Other Names: Procoralan
  Arms: ivabradine (add-on)

SUMMARY:
MODIfY is a prospective, single center, open label, randomized, controlled two arms, Phase II-trial to evaluate the ability of ivabradine to reduce an elevated heart rate in Multiple Organ Dysfunction Syndrome (MODS) patients. The primary end point is the proportion of patients with a reduction of heart rate by at least 10 beats per minute (bpm) within 4 days. This trial will randomize 70 patients (men and women, aged ≥ 18 years) with newly diagnosed MODS (Acute Physiology and Chronic Health Evaluation (APACHE) II-score ≥ 20, diagnosis within ≤ 24 hours), with an elevated heart rate (sinus rhythm with HR ≥ 90 bpm) and contraindications to beta-blockers (BBs). Treatment period will last 4 days. All patients will be followed for up to six months.

DETAILED DESCRIPTION:
Background: Heart rate (HR) is of relevant prognostic value not only in the general population and patients with cardiovascular disease but also in critically ill patients with multiple organ dysfunction syndrome (MODS). A raised heart rate in MODS patients is associated with a worse prognosis. Beta-blocker (BB) administration showed to improve autonomic function and exhibited a significantly reduced mortality in MODS. In most cases negative inotropic effects prevent administration of BB in MODS patients which often are treated with catecholamines. In this trial we investigate, whether the "funny current" (If) inhibitor ivabradine is able to reduce pathologically elevated heart rate in MODS- patients.

The investigators hypothesized that critically ill patients could derive particular benefit from the specific HR-lowering agent ivabradine.

Methods: MODIfY is a prospective, single center, open label, randomized, controlled two arms, Phase II-trial to evaluate the ability of ivabradine to reduce an elevated heart rate in MODS patients. The primary end point is the proportion of patients with a reduction of heart rate by at least 10 beats per minute (bpm) within 4 days. This trial will randomize 70 patients (men and women, aged ≥18 years) with newly diagnosed MODS (Acute Physiology and Chronic Health Evaluation (APACHE) II-score ≥20, diagnosis within ≤24 hours), with an elevated heart rate (sinus rhythm with HR ≥90 bpm) and contraindications to BBs. Treatment period will last 4 days. All patients will be followed for up to six months.

ELIGIBILITY:
Inclusion Criteria:

* Multiple organ dysfunction syndrome (APACHE II score ≥ 20) due to coronary and non-coronary etiology
* Multiple organ dysfunction syndrome diagnosed ≤ 24 h
* Sinus rhythm with heart rate ≥ 90bpm
* Existing contraindications to beta-receptor blockade
* Written informed consent or identified or suspected positive will with respect to the trial treatment

Exclusion Criteria:

* Patients who have not yet completed the 18th year of age
* Pregnancy, lactation
* Patients with a history of pre-existing chronic renal failure with a glomerular filtration rate <30ml/min
* Patients with malignant hyperthermia
* Burn patients
* Patients with acute rejection after organ transplantation
* Patients with bleedings and need for transfusion
* Resuscitated patients with suspected hypoxic brain injury
* Patients who have participated or participate in other studies within the last 3 months
* Other types of shock than septic or cardiogenic shock
* Patients with severe valvular heart disease
* Hypersensitivity to the active substance or any of the excipients
* Severe hepatic insufficiency
* Sick sinus syndrome
* Sinu-atrial block
* pacemaker-dependency
* 3rd degree AV block
* Use of potent cytochrome P450 3A4 inhibitors such as antifungals of the azole -type (ketoconazole, itraconazole), macrolide antibiotics (clarithromycin, erythromycin per os, josamycin, telithromycin), HIV protease inhibitors (nelfinavir, ritonavir) and nefazodone (see Summary of Product Characteristics (SPC))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-11 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
mean heart rate | 4 days
  percenage of patients with a reduction of the mean heart rate of at least 10 bpm 96 hours after the start of trial treatment

SECONDARY OUTCOMES:
morbidity | 4 days
  group-differences and patient-related changes of morbidity measured by serial APACHE II score monitoring and Sequential Organ Failure Assessment (SOFA) score monitoring
hemodynamic parameters | 4 days
  group-differences and patient-related changes of hemodynamic parameters (cardiac index and cardiac power index) as a consequence of ivabradine treatment
catecholamine dosage | 4 days
  required catecholamine dosage measured by a vasopressor score
microcirculation | 4 days
  improvement of microcirculation as measured by sublingual capillary density and flow
endothelial function | 4 days
  improvement of endothelial function as measured by the "Reactive hyperemia peripheral arterial tonometry-index"
mean heart rate | 48 hours
  comparison of the mean heart rate between the treatment and control group after 24 and 48 hours
mortality | 6 months
  28-day and 6 months mortality
cardiac autonomic dysfunction | 4 days
  impact on cardiac autonomic dysfunction (heart rate variability quantified by time domain measurements (standard deviation of normal to normal interval (SDNN)) and frequency domain measurements (very low frequency (VLF)-, high frequency (HF)- and low frequency (LF)-power) as well as minimum, maximum, day and night heart rate)
number of participants with adverse events as a measure of safety and tolerability | 6 months
plasma levels of ivabradine in patients with MODS | 4 days
  daily measurement of plasma levels during the treatment period (4 days)
Differences of mortality in different age groups and MODS groups | 6 months
  age sub-groups:
  1. patients <70 years on day of inclusion
  2. patients ≥70 years on day of inclusion
  MODS sub-groups:
  1. patients with cardiogenic MODS
  2. patients with septic MODS
Differences of adverse events in different age groups and MODS groups | 6 months
  age sub-groups:
  1. patients <70 years on day of inclusion
  2. patients ≥70 years on day of inclusion
  MODS sub-groups:
  1. patients with cardiogenic MODS
  2. patients with septic MODS
Differences of heart rate in different age groups and MODS groups | 6 months
  age sub-groups:
  1. patients <70 years on day of inclusion
  2. patients ≥70 years on day of inclusion
  MODS sub-groups:
  1. patients with cardiogenic MODS
  2. patients with septic MODS

CONTACTS AND LOCATIONS:
Overall Officials: Karl Werdan, MD, Professor, Study Chair — Medical Faculty of the Martin-Luther-University Halle-Wittenberg, Germany; Henning Ebelt, MD, Principal Investigator — Medical Faculty of the Martin-Luther-University Halle-Wittenberg, Germany; Sebastian Nuding, MD, Principal Investigator — Medical Faculty of the Martin-Luther-University Halle-Wittenberg, Germany
Locations (1):
- Department of Medicine III of the University Clinics Halle (Saale) of the Martin-Luther-University Halle-Wittenberg, Halle, Saxony-Anhalt, Germany

REFERENCES:
- [Background] Borer JS. Drug insight: If inhibitors as specific heart-rate-reducing agents. Nat Clin Pract Cardiovasc Med. 2004 Dec;1(2):103-9. doi: 10.1038/ncpcardio0052. PMID 16265314
- [Background] American College of Chest Physicians/Society of Critical Care Medicine Consensus Conference: definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. Crit Care Med. 1992 Jun;20(6):864-74. PMID 1597042
- [Background] Bernard GR, Vincent JL, Laterre PF, LaRosa SP, Dhainaut JF, Lopez-Rodriguez A, Steingrub JS, Garber GE, Helterbrand JD, Ely EW, Fisher CJ Jr; Recombinant human protein C Worldwide Evaluation in Severe Sepsis (PROWESS) study group. Efficacy and safety of recombinant human activated protein C for severe sepsis. N Engl J Med. 2001 Mar 8;344(10):699-709. doi: 10.1056/NEJM200103083441001. PMID 11236773
- [Background] Bernardin G, Strosberg AD, Bernard A, Mattei M, Marullo S. Beta-adrenergic receptor-dependent and -independent stimulation of adenylate cyclase is impaired during severe sepsis in humans. Intensive Care Med. 1998 Dec;24(12):1315-22. doi: 10.1007/s001340050768. PMID 9885886
- [Background] Cooney MT, Vartiainen E, Laatikainen T, Juolevi A, Dudina A, Graham IM. Elevated resting heart rate is an independent risk factor for cardiovascular disease in healthy men and women. Am Heart J. 2010 Apr;159(4):612-619.e3. doi: 10.1016/j.ahj.2009.12.029. PMID 20362720
- [Background] Cucherat M. Quantitative relationship between resting heart rate reduction and magnitude of clinical benefits in post-myocardial infarction: a meta-regression of randomized clinical trials. Eur Heart J. 2007 Dec;28(24):3012-9. doi: 10.1093/eurheartj/ehm489. Epub 2007 Nov 2. PMID 17981830
- [Background] Heidland UE, Strauer BE. Left ventricular muscle mass and elevated heart rate are associated with coronary plaque disruption. Circulation. 2001 Sep 25;104(13):1477-82. doi: 10.1161/hc3801.096325. PMID 11571239
- [Background] Hennen R, Friedrich I, Hoyer D, Nuding S, Rauchhaus M, Schulze M, Schlisske S, Schwesig R, Schlitt A, Buerke M, Muller-Werdan U, Werdan K, Schmidt H. [Autonomic dysfunction and beta-adrenergic blockers in multiple organ dysfunction syndrome]. Dtsch Med Wochenschr. 2008 Nov;133(48):2500-4. doi: 10.1055/s-0028-1100944. Epub 2008 Nov 19. German. PMID 19021079
- [Background] Herndon DN, Barrow RE, Rutan TC, Minifee P, Jahoor F, Wolfe RR. Effect of propranolol administration on hemodynamic and metabolic responses of burned pediatric patients. Ann Surg. 1988 Oct;208(4):484-92. doi: 10.1097/00000658-198810000-00010. PMID 3052328
- [Background] Herndon DN, Hart DW, Wolf SE, Chinkes DL, Wolfe RR. Reversal of catabolism by beta-blockade after severe burns. N Engl J Med. 2001 Oct 25;345(17):1223-9. doi: 10.1056/NEJMoa010342. PMID 11680441
- [Background] Kjekshus J. Heart rate reduction--a mechanism of benefit? Eur Heart J. 1987 Dec;8 Suppl L:115-22. doi: 10.1093/eurheartj/8.suppl_l.115. No abstract available. PMID 2897914
- [Background] Kjekshus JK. Importance of heart rate in determining beta-blocker efficacy in acute and long-term acute myocardial infarction intervention trials. Am J Cardiol. 1986 Apr 25;57(12):43F-49F. doi: 10.1016/0002-9149(86)90888-x. PMID 2871745
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Background] Levy MM, Fink MP, Marshall JC, Abraham E, Angus D, Cook D, Cohen J, Opal SM, Vincent JL, Ramsay G; International Sepsis Definitions Conference. 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference. Intensive Care Med. 2003 Apr;29(4):530-8. doi: 10.1007/s00134-003-1662-x. Epub 2003 Mar 28. PMID 12664219
- [Background] Manz M, Reuter M, Lauck G, Omran H, Jung W. A single intravenous dose of ivabradine, a novel I(f) inhibitor, lowers heart rate but does not depress left ventricular function in patients with left ventricular dysfunction. Cardiology. 2003;100(3):149-55. doi: 10.1159/000073933. PMID 14631136
- [Background] Marshall JC, Cook DJ, Christou NV, Bernard GR, Sprung CL, Sibbald WJ. Multiple organ dysfunction score: a reliable descriptor of a complex clinical outcome. Crit Care Med. 1995 Oct;23(10):1638-52. doi: 10.1097/00003246-199510000-00007. PMID 7587228
- [Background] Muller-Werdan U, Buerke M, Ebelt H, Heinroth KM, Herklotz A, Loppnow H, Russ M, Schlegel F, Schlitt A, Schmidt HB, Soffker G, Werdan K. Septic cardiomyopathy - A not yet discovered cardiomyopathy? Exp Clin Cardiol. 2006 Fall;11(3):226-36. PMID 18651035
- [Background] Norbury WB, Jeschke MG, Herndon DN. Metabolism modulators in sepsis: propranolol. Crit Care Med. 2007 Sep;35(9 Suppl):S616-20. doi: 10.1097/01.CCM.0000278599.30298.80. PMID 17713418
- [Background] Opal S, Laterre PF, Abraham E, Francois B, Wittebole X, Lowry S, Dhainaut JF, Warren B, Dugernier T, Lopez A, Sanchez M, Demeyer I, Jauregui L, Lorente JA, McGee W, Reinhart K, Kljucar S, Souza S, Pribble J; Controlled Mortality Trial of Platelet-Activating Factor Acetylhydrolase in Severe Sepsis Investigators. Recombinant human platelet-activating factor acetylhydrolase for treatment of severe sepsis: results of a phase III, multicenter, randomized, double-blind, placebo-controlled, clinical trial. Crit Care Med. 2004 Feb;32(2):332-41. doi: 10.1097/01.CCM.0000108867.87890.6D. PMID 14758145
- [Background] Palatini P, Julius S. Association of tachycardia with morbidity and mortality: pathophysiological considerations. J Hum Hypertens. 1997 Aug;11 Suppl 1:S19-27. PMID 9321736
- [Background] Pilz G, Appel R, Kreuzer E, Werdan K. Comparison of early IgM-enriched immunoglobulin vs polyvalent IgG administration in score-identified postcardiac surgical patients at high risk for sepsis. Chest. 1997 Feb;111(2):419-26. doi: 10.1378/chest.111.2.419. PMID 9041991
- [Background] Pilz G, Kaab S, Kreuzer E, Werdan K. Evaluation of definitions and parameters for sepsis assessment in patients after cardiac surgery. Infection. 1994 Jan-Feb;22(1):8-17. doi: 10.1007/BF01780757. PMID 8181848
- [Background] Pilz G, Werdan K. Cardiovascular parameters and scoring systems in the evaluation of response to therapy in sepsis and septic shock. Infection. 1990 Sep-Oct;18(5):253-62. doi: 10.1007/BF01646996. PMID 2276817
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Schmidt H, Muller-Werdan U, Hoffmann T, Francis DP, Piepoli MF, Rauchhaus M, Prondzinsky R, Loppnow H, Buerke M, Hoyer D, Werdan K. Autonomic dysfunction predicts mortality in patients with multiple organ dysfunction syndrome of different age groups. Crit Care Med. 2005 Sep;33(9):1994-2002. doi: 10.1097/01.ccm.0000178181.91250.99. PMID 16148471
- [Background] Schmidt HB, Werdan K, Muller-Werdan U. Autonomic dysfunction in the ICU patient. Curr Opin Crit Care. 2001 Oct;7(5):314-22. doi: 10.1097/00075198-200110000-00002. PMID 11805528
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Thollon C, Cambarrat C, Vian J, Prost JF, Peglion JL, Vilaine JP. Electrophysiological effects of S 16257, a novel sino-atrial node modulator, on rabbit and guinea-pig cardiac preparations: comparison with UL-FS 49. Br J Pharmacol. 1994 May;112(1):37-42. doi: 10.1111/j.1476-5381.1994.tb13025.x. PMID 8032660
- [Background] Vincent JL, Angus DC, Artigas A, Kalil A, Basson BR, Jamal HH, Johnson G 3rd, Bernard GR; Recombinant Human Activated Protein C Worldwide Evaluation in Severe Sepsis (PROWESS) Study Group. Effects of drotrecogin alfa (activated) on organ dysfunction in the PROWESS trial. Crit Care Med. 2003 Mar;31(3):834-40. doi: 10.1097/01.CCM.0000051515.56179.E1. PMID 12626993
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Werdan K, Pilz G, Bujdoso O, Fraunberger P, Neeser G, Schmieder RE, Viell B, Marget W, Seewald M, Walger P, Stuttmann R, Speichermann N, Peckelsen C, Kurowski V, Osterhues HH, Verner L, Neumann R, Muller-Werdan U; Score-Based Immunoglobulin Therapy of Sepsis (SBITS) Study Group. Score-based immunoglobulin G therapy of patients with sepsis: the SBITS study. Crit Care Med. 2007 Dec;35(12):2693-2701. PMID 18074471
- [Background] Werdan K, Schmidt H, Ebelt H, Zorn-Pauly K, Koidl B, Hoke RS, Heinroth K, Muller-Werdan U. Impaired regulation of cardiac function in sepsis, SIRS, and MODS. Can J Physiol Pharmacol. 2009 Apr;87(4):266-74. doi: 10.1139/Y09-012. PMID 19370080
- [Background] Wilhelmsen L, Berglund G, Elmfeldt D, Tibblin G, Wedel H, Pennert K, Vedin A, Wilhelmsson C, Werko L. The multifactor primary prevention trial in Goteborg, Sweden. Eur Heart J. 1986 Apr;7(4):279-88. doi: 10.1093/oxfordjournals.eurheartj.a062065. PMID 3720755
- [Background] Zorn-Pauly K, Pelzmann B, Lang P, Machler H, Schmidt H, Ebelt H, Werdan K, Koidl B, Muller-Werdan U. Endotoxin impairs the human pacemaker current If. Shock. 2007 Dec;28(6):655-661. PMID 18092381
- [Background] Zuppa AF, Nadkarni V, Davis L, Adamson PC, Helfaer MA, Elliott MR, Abrams J, Durbin D. The effect of a thyroid hormone infusion on vasopressor support in critically ill children with cessation of neurologic function. Crit Care Med. 2004 Nov;32(11):2318-22. doi: 10.1097/01.ccm.0000146133.52982.17. PMID 15640648
- [Derived] Nuding S, Ebelt H, Hoke RS, Krummenerl A, Wienke A, Muller-Werdan U, Werdan K. Reducing elevated heart rate in patients with multiple organ dysfunction syndrome by the I (f) (funny channel current) inhibitor ivabradine : MODI (f)Y trial. Clin Res Cardiol. 2011 Oct;100(10):915-23. doi: 10.1007/s00392-011-0323-2. Epub 2011 Jun 3. PMID 21638157